CLINICAL TRIAL: NCT03146403
Title: A Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy and Safety of a Maintenance Dose of GEN-003 in Subjects With Genital Herpes Infection
Brief Title: Maintenance Dose Study of GEN-003 in Subjects With Genital Herpes Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 2017 business decision to cease GEN-003 spending.
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-003-005
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Genital Herpes; HSV-2 Infection
Keywords: HSV; Herpes; Genital Herpes; Vaccine
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — M2 protein, Influenza A virus; Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GEN-003 (Experimental): 60μg of each GEN-003 antigen with 50μg Matrix-M2 adjuvant, administered as a 0.5mL intramuscular (IM) injection
  Interventions: Biological: GEN-003; Biological: Matrix-M2
- Placebo (Placebo Comparator): 0.9% normal saline administered as a 0.5mL intramuscular (IM) injection
  Interventions: Other: 0.9% normal saline

INTERVENTIONS:
Biological: GEN-003 — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP4 and glycoprotein D
  Other Names: HSV Therapeutic Vaccine
  Arms: GEN-003
Biological: Matrix-M2 — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: Adjuvant
  Arms: GEN-003
Other: 0.9% normal saline — Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this clinical study is to see if a maintenance dose of GEN-003 reduces the number of days that subjects have a genital herpes recurrence. The second purpose of the study is to evaluate the safety and tolerability of a maintenance dose of GEN-003.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial of GEN-003 in subjects who have received previous doses of GEN-003 in the GEN-003-003 clinical trial. Eligible subjects will be randomized in a 1:1 ratio to receive 1 intramuscular (IM) dose (the maintenance dose) of GEN-003 or placebo.

Subjects will use a daily electronic reporting tool for reporting the presence or absence of genital herpes lesions, and severity of genital herpes symptoms.

GEN-003-005 was originally designed to follow subjects for 12 months after the maintenance dose but a business decision, unrelated to product safety, was made by Genocea Biosciences in 3Q2017 to cease GEN-003 spending and activities.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study GEN-003-003
* Received all 3 GEN-003 doses (any dose combination) in Study GEN-003-003
* Received last dose of GEN-003 within 11 to 18 months prior
* Reported data in the daily electronic reporting period on at least 80% of days in Study GEN-003-003
* Collected at least 45 swabs (of 56 total expected swabs) during the Month 11 to 12 swab collection period in Study GEN-003-003
* Willing and able to provide written informed consent
* Willing to perform and comply with all study procedures
* Postmenopausal or willing to practice a highly effective method of contraception for 28 days before and 90 days after enrollment

Exclusion Criteria:

* Did not meet all eligibility criteria in Study GEN-003-003, or received incorrect treatment in Study GEN-003-003
* Use of suppressive antiviral medication within 14 days prior
* Use of topical steroids or antiviral medication in the anogenital region within 14 days prior
* Use of tenofovir, lysine, or other medication or supplement known or purported to affect HSV recurrence frequency or intensity within 14 days prior
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or herpes meningitis or encephalitis
* Immunocompromised individuals
* Diagnosis or suspicion of an AESI
* Diagnosis or suspicion of any other autoimmune disease not listed in Appendix 4 of the protocol
* Vaccine-related SAE in GEN-003-003
* Known current infection with HIV or hepatitis B or C virus
* History of hypersensitivity to any component of the vaccine
* Prior receipt of another vaccine containing HSV-2 antigens other than GEN-003
* Receipt of any IP within 30 days prior to the maintenance dose of GEN-003/placebo
* Receipt of any blood product within 90 days prior to the maintenance dose
* Receipt of a live vaccine within 28 days prior to or any other vaccine within 14 days prior to maintenance dose
* Planned use of any vaccine from the maintenance dose to 28 days after the maintenance dose
* Pregnant or nursing women
* History of drug or alcohol abuse
* Other active, uncontrolled comorbidities
* Changes to medication used to manage an underlying comorbidity within 60 days prior

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - UNC Health, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - NW Dermatology and Research Clinic, Portland, Oregon
  - Tekton Research, Austin, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GEN-003 | Placebo
Started | 16 | 17
Completed | 14 | 14
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GEN-003 | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Full Range); unit: years] | 39.9 [27 to 50] | 40.2 [30 to 52] | 40.1 [27 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33
Weight [Mean (Full Range); unit: kilograms] | 82.34 [54.0 to 140.5] | 79.20 [53.5 to 119.3] | 80.72 [53.5 to 140.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With Genital Herpes Lesions
Description: Subject-reported via electronic diary
Time Frame: The 6-month period after vaccination
Population: Results for the placebo group are based on 16 subjects, after excluding one subject who reported no electronic diary lesion data.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | GEN-003 | Placebo
Number analyzed (Participants) | 16 | 16
percentage of days | 2.58 [0.0 to 21.8] | 4.23 [0.0 to 13.5]
Statistical Analysis 1: Comparison: GEN-003 vs Placebo; Test type: Superiority; p = 0.7474, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Genital Herpes Recurrences
Description: Subject-reported via electronic diary
Time Frame: The 6-month period after vaccination
Population: as for outcome 1
Measure: Median (Full Range); unit: recurrences
Arm/Group | GEN-003 | Placebo
Number analyzed (Participants) | 16 | 16
recurrences | 1.50 [0.0 to 6.0] | 1.50 [0.0 to 9.0]
Statistical Analysis 1: Comparison: GEN-003 vs Placebo; Test type: Superiority; p = 0.6450, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Subjects Without Genital Herpes Recurrence
Description: Subject-reported via electronic diary
Time Frame: 6 months after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GEN-003 | Placebo
Number analyzed (Participants) | 16 | 16
Participants
  No Recurrence | 1 | 3
  With Recurrence | 13 | 12
  Unknown | 2 | 1
Statistical Analysis 1: Comparison: GEN-003 vs Placebo; Test type: Superiority; p = 0.3157, Chi-squared

4. Secondary Outcome: Days Until First Genital Herpes Recurrence
Description: Subject-reported via electronic diary
Time Frame: The 6-month period after vaccination
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | GEN-003 | Placebo
Number analyzed (Participants) | 16 | 16
days | 25 [6.0 to 85.0] | 51 [17.0 to 116.0]
Statistical Analysis 1: Comparison: GEN-003 vs Placebo; Test type: Superiority; p = 0.3869, Log Rank

5. Secondary Outcome: Duration of Genital Herpes Recurrences
Description: Time in days per genital herpes recurrence
Time Frame: The 6-month period after vaccination
Measure: Median (Full Range); unit: days
Arm/Group | GEN-003 | Placebo
Number analyzed (Participants) | 13 | 12
days | 2.83 [1 to 7] | 3.40 [1 to 6]
Statistical Analysis 1: Comparison: GEN-003 vs Placebo; Test type: Superiority; p = 0.2200, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events were systematically collected for 7 days after the maintenance dose. AEs were recorded for 12 months of followup after the maintenance dose administration.
Description: Systematic AE results for the placebo group are based on 16 subjects since one subject who withdrew from the study did not report local reactions and systemic events data.
Arm/Group | GEN-003 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 16/16 | 10/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GEN-003 (N=16) | Placebo (N=17)
Fatigue (General disorders) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Disturbance in attention (General disorders) | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 1 | 0
Injection Site Pain (General disorders) | 15 | 3/16
Injection Site Tenderness (General disorders) | 15 | 7/16
Injection Site Swelling (General disorders) | 13 | 3/16
Injection Site Redness (General disorders) | 5 | 2/16
Fever (General disorders) | 3 | 0/16 — ≥100.4°F
Headache (Nervous system disorders) | 13 | 7/16
Chills (General disorders) | 10 | 1/16
Fatigue (General disorders) | 14 | 5/16
Nausea (Gastrointestinal disorders) | 6 | 1/16
Diarrhea (Gastrointestinal disorders) | 3 | 1/16
Muscle Aches (Musculoskeletal and connective tissue disorders) | 15 | 2/16

LIMITATIONS AND CAVEATS:
Small numbers of enrolled subjects likely led to a lack of statistical power. After a 2017 business decision to cease GEN-003 spending, the outcome measures were reduced to 6 months of follow up, rather than the originally planned 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT03146403/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03146403/SAP_001.pdf